CLINICAL TRIAL: NCT04962958
Title: Prospective, Single-arm, Multicenter Clinical Study of Hepatic Artery Infusion Chemotherapy With Donafenib for Adjuvant Treatment of HCC Patients With High Risk of Recurrence After Hepatectomy.
Brief Title: Hepatic Artery Infusion Chemotherapy Plus Donafenib in Patients With Hepatocellular Carcinoma After Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Meng Chao Hepatobiliary Hospital of Fujian Medical University (Other); Huashan Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-KY-047
Record Dates: First submitted 2021-07-06; First posted 2021-07-15 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Carcinoma; Carcinoma, Hepatocellular; Liver Neoplasms; Digestive System Neoplasms; Antineoplastic Agents; Donafenib; Fluorouracil; Oxaliplatin; Antimetabolites
Keywords: Hepatocellular Carcinoma; Hepatic arterial infusion chemotherapy; Donafenib
MeSH Terms: conditions — Carcinoma; Carcinoma, Hepatocellular; Liver Neoplasms; Digestive System Neoplasms | interventions — Folfox protocol; Oxaliplatin; Fluorouracil; Leucovorin; donafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC+Donafenib (Experimental): Donafenib combined with Hepatic arterial infusion chemotherapy with Folfox Protocol
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Folfox Protocol; Drug: Donafenib

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — administration of Oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
  Other Names: HAIC
Drug: Folfox Protocol — Oxaliplatin , fluorouracil, and leucovorin
  Other Names: Oxaliplatin , fluorouracil, and leucovorin
Drug: Donafenib — administration of Donafenib

SUMMARY:
This is an open-label，multi-center ，non-randomized ，single arm exploratory study . This clinical study is an investigator-initiated clinical trial（IIT ）. The objective of this study is to evaluate if the addition of hepatic artery infusion chemotherapy (HAIC) and Donafenib after curative resection for hepatocellular carcinoma patients with a solitary tumor≥5 cm and microvascular invasion （MVI） will prevent or delay the recurrence of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, male or female;
2. Naive patients with hepatocellular carcinoma pathologically diagnosed who have Underwent radical hepatectomy 4-8 weeks before enrollment;
3. HCC patients with a solitary tumor≥5 cm and Microvascular invasion;
4. Child-Pugh score A/B(≤7);
5. ECOG PS score 0-1;
6. No residual tumor lesions were confirmed on imaging more than 4 weeks after surgery;
7. The main organ functions meet the following criteria within 14 days before enrollment; (1)Hemoglobin(HB)≥100 g/L (2)neutrophils(ANC)≥1.5×10^9 /L, (3)platelet count(PLT)≥75×10^9/L; (4)ALB≥28g/L (5)alanine aminotransferase(ALT), aspartate aminotransferase(AST)<5×ULN (6)Total bilirubin (TBIL)<1.5×ULN (7)Plasma creatinine ≤1.5×ULN with a creatinine clearance≥50mL/min (8)Activation Partial Thrombin Activation Time (APTT) and International Normalized Ratio (INR)≤1.5×ULN
8. Subjects voluntarily enrolled in the study, signed an informed consent form, followed well and cooperated with the follow-up

Exclusion Criteria:

1. Patients who have received any hepatocellular carcinoma-related systemic therapy before enrollment; including targeted therapy such as sorafenib, lenvatinib, and regorafenib, or immunomodulators such as anti-PD-1, anti-PD-L1, and anti-CTLA-4 Treatment, excluding antiviral treatment; if the patient has used traditional Chinese medicine with anti-tumor indications, it must be> 2 weeks or 5 drug half-lives (whichever is longer). Patients whose adverse events caused by treatment have not recovered to ≤ CTCAE Grade 1;
2. Patients who have received other adjuvant treatments (except antiviral therapy) after radical hepatectomy, including adjuvant local treatments (such as transarterial chemoembolization [TACE]);
3. Hepatic veins, portal veins, bile ducts, or inferior vena cava can be visually or microscopically seen with tumor thrombi
4. Diagnosed with lymph node invasion or extrahepatic metastasis;
5. Number of tumors≥2;
6. A history of other malignant tumours within the last five years, except for cured skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ or other carcinoma in situ;
7. Pregnant or breastfeeding women; males or females of childbearing age who are unwilling or unable to take effective contraceptive measures
8. Known history of alcohol, psychotropic drug or other drug abuse within 6 months before entry into the study 9.Those the researcher deems inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
2-year cumulative recurrence-free survival rate | 2-year
  This is defined as the length of time (days) that the patient survives since study registration without any signs or symptoms of locoregional HCC assessed by structured clinical and radiological (clinical) follow-up . If at close-out date of the study, there are no signs of locoregional recurrence, the patient will be censored to the date of the most recent follow-up examination. The 2-year cumulative incidence rates will be estimated from the curves and its associated 95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
1-year recurrence-free survival rate | 1-year
  This is defined as the length of time (days) that the patient survives since study registration without any signs or symptoms of locoregional HCC assessed by structured clinical and radiological (clinical) follow-up . If at close-out date of the study, there are no signs of locoregional recurrence, the patient will be censored to the date of the most recent follow-up examination. The 1-year cumulative incidence rates will be estimated from the curves and its associated 95% confidence intervals will be calculated.
Disease-free survival | 2-year
  from the date of enrollment to tumor recurrence or Death
Overall Survival | approximately 60 months from first patient first visit
  from the date of enrollment to Death
Adverse Events | 30 days
  Number of adverse events. Postoperative adverse events were graded based on CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, PHD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Lei Zhang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No